CLINICAL TRIAL: NCT05110235
Title: PERCUTANEOUS ENDOSCOPIC GASTROSTOMY APPLICATION EXPERIENCES TO GERIATRIC PATIENTS IN PALLIATIVE CARE UNIT
Brief Title: PEG Application Experiences to Geriatric Patients
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Murat Ferhat Ferhatoglu, Medical Doctor, Assistant Professor, Principal investigator, Okan University
Other Study IDs: 56665618-204.01.08
Record Dates: First submitted 2021-10-13; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Nutrient Deficiency; Gastrostomy
Keywords: Geriatrics; Nutrition; PEG; Gastrostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Percutaneous endoscopic gastrostomy (PEG) is currently the chosen minimally invasive, endoscopic procedure for medium- and long-term enteral feeding in cases who need palliative care. The presented study evaluated geriatric (> 65-year-old) PEG-applied patients at our institution.

DETAILED DESCRIPTION:
Palliative care is a treatment method that focuses on the patient and patient's family, aims to minimize the complaints caused by chronic diseases that cannot be treated, and increases life quality. The National Institute for Health and Care Excellence defines palliative care as; the active, holistic care of patients with an advanced progressive illness. Management of pain and other symptoms and providing psychological, social, and spiritual support is paramount. Anorexia, weight loss, and sarcopenia are highly visible and distressing reminders of the life-limiting disease's influence on patients who require palliative care. Given this multifaceted and significant role, it is not unexpected that nutritional treatment method choices can be challenging.

Percutaneous endoscopic gastrostomy (PEG) is a minimally-invasive endoscopic procedure that creates a passage from the patient's stomach to the abdominal wall via a feeding tube and provides a means of feeding if oral intake is not adequate. This safe and effective minimally-invasive option has been utilized in medical practice for over 40 years. PEG has advantages such as being minimally invasive, causing a low rate of complications and morbidity, and providing a long-lasting and safe feeding route. It is currently the chosen procedure for medium- and long-term enteral feeding in cases who need palliative care.

The application of PEG in geriatric-palliative care has not been well discussed. With the development of endoscopic procedures and PEG devices, this minimally invasive method can be applied more safely, even in challenging cases. This study discuss the indications of PEG in the field of palliative care of geriatric patients.

ELIGIBILITY:
Inclusion Criteria: PEG applied >65-year-old patients at our institution between December 2017 and March 2021 -

Exclusion Criteria: We excluded the patients who were not treated in our palliative care center

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We retrospectively assessed the medical datum of PEG applied >65-year-old patients at our institution between December 2017 and March 2021. And, we excluded the patients who were not treated in our palliative care center. Table 1. shows the contraindications for PEG placement.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (gr/dl) | 30 days
  30 th day hemoglobin levels after PEG application
Albumin (gr/dl) | 30 days
  30 th day albumin levels after PEG application

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University Hospital, Istanbul, Turkey (Türkiye)